CLINICAL TRIAL: NCT02981498
Title: Phase II Trial of Sorafenib Combined With Concurrent Hepatic Arterial Infusion (HAI) of Oxaliplatin, 5-fluorouracil and Leucovorin for Hepatocellular Carcinoma
Brief Title: Phase II Trial of Sorafenib Combined With Concurrent HAIC for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Shi Ming, Proffesor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S027
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatic arterial infusion chemotherapy; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib combined with HAIC (Experimental): Sorafenib combined with Hepatic arterial infusion chemotherapy with Folfox Protocol
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Folfox Protocol

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of Oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries
Drug: Folfox Protocol — Oxaliplatin , fluorouracil, and leucovorin

SUMMARY:
To evaluate safety and efficacy of combined hepatic arterial infusion (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin and sorafenib in patients with advanced hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
In most current guidelines, unresectable HCC with major PVTT are considered not generally suitable for transarterial chemoembolization, and sorafenib is recommended as standard care.3-5 However, for patients with major PVTT, the median overall survival of those treated with sorafenib monotherapy was only 3.1 to 6.0 months.

Whether combining sorafenib with hepatic arterial infusion (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin is safe, well tolerated, and efficacious remains unknown, with no prospective clinical data currently available.The investigators therefore conducted a prospective single center, single-arm phase II trial to evaluate the safety and efficacy of sorafenib combined with HAIC in patients with unresectable advanced HCC.

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* diagnosed with major or main portal vein invasion (Vp3 or Vp4)
* KPS≥70；
* with no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

  * Platelet count ≥ 75,000/µL
  * Hemoglobin ≥ 8.5 g/dL
  * Total bilirubin ≤ 30mmol/L
  * Serum albumin ≥ 30 g/L
  * ASL and AST ≤ 5 x upper limit of normal
  * Serum creatinine ≤ 1.5 x upper limit of normal
  * INR ≤ 1.5 or PT/APTT within normal limits
  * Absolute neutrophil count (ANC) >1,500/mm3
* Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug
* Serious non-healing wound, ulcer, or bone fracture
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
progression-free survival rate | 3 month

SECONDARY OUTCOMES:
Objective response | 3 month
OS | 12 months
  Overall Survival
AE event | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ming Shi, MD, Principal Investigator — The Department of Hepatobiliary Oncology of Sun Yat-sen University Cancer Center
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Result] Ando E, Yamashita F, Tanaka M, Tanikawa K. A novel chemotherapy for advanced hepatocellular carcinoma with tumor thrombosis of the main trunk of the portal vein. Cancer. 1997 May 15;79(10):1890-6. doi: 10.1002/(sici)1097-0142(19970515)79:103.0.co;2-k. PMID 9149014
- [Result] Luo J, Guo RP, Lai EC, Zhang YJ, Lau WY, Chen MS, Shi M. Transarterial chemoembolization for unresectable hepatocellular carcinoma with portal vein tumor thrombosis: a prospective comparative study. Ann Surg Oncol. 2011 Feb;18(2):413-20. doi: 10.1245/s10434-010-1321-8. Epub 2010 Sep 14. PMID 20839057
- [Derived] He MK, Zou RH, Li QJ, Zhou ZG, Shen JX, Zhang YF, Yu ZS, Xu L, Shi M. Phase II Study of Sorafenib Combined with Concurrent Hepatic Arterial Infusion of Oxaliplatin, 5-Fluorouracil and Leucovorin for Unresectable Hepatocellular Carcinoma with Major Portal Vein Thrombosis. Cardiovasc Intervent Radiol. 2018 May;41(5):734-743. doi: 10.1007/s00270-017-1874-z. Epub 2018 Jan 11. PMID 29327075